CLINICAL TRIAL: NCT03332056
Title: The Use of Belladonna and Opium (B&O) Suppository in the Treatment of Postoperative Stent Pain: A Randomized, Double-Blinded Control Study
Brief Title: The Use of Belladonna and Opium Suppository in the Treatment of Postoperative Stent Pain
Acronym: B&O
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jonathan Harper, MD, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 44862
Record Dates: First submitted 2015-11-04; First posted 2017-11-06 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Nephrolithiasis
Keywords: Ureteral stent pain; nephrolithiasis; kidney stone
MeSH Terms: conditions — Nephrolithiasis; Kidney Calculi | interventions — Opium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Belladonna and Opium (B&O) suppository (Active Comparator): A single belladonna and opium suppository, dose-weight calculated, administered immediately following patient positioning prior to instrumentation. The pharmacologically active ingredients that are present in the belladonna extract consist of atropine and scopolamine. Opium is compound drug that is composed of 20 alkaloids. The principle alkaloid that derives the majority of its effect is its morphine content and acts as a narcotic analgesic by increasing the pain threshold or the magnitude of stimulus required to evoke pain.
  Interventions: Drug: Belladonna and Opium
- Placebo Suppository (Placebo Comparator): placebo suppository
  Interventions: Other: Placebo suppository

INTERVENTIONS:
Drug: Belladonna and Opium
  Other Names: B&O
  Arms: Belladonna and Opium (B&O) suppository
Other: Placebo suppository
  Arms: Placebo Suppository

SUMMARY:
The purpose of this study is to determine if preemptive B&O suppository placement will decrease post-operative pain in patients undergoing ureteral stent placement.

DETAILED DESCRIPTION:
Purpose: Nephrolithiasis has an incidence of 10-15% in the US with 66% of practicing urologists placing a ureteral stent after each procedure. Ureteral stents are commonly placed to prevent or alleviate ureteral obstruction and ureteral stents are not well tolerated with up to 80% of patients reporting stent discomfort. These symptoms include urinary frequency, urgency, dysuria and incomplete emptying. Patients also frequently report suprapubic pain, hematuria and incontinence. Ureteral stents are placed either alone or in conjunction with other surgeries where ureteral access is obtained.

To date, however, there is no convincing data that altering stent characteristics or the use of a single drug dramatically improves stent discomfort for patients. Prior studies on oral therapies including alpha blockers and anti-muscarinics have shown some promise in improving stent comfort, however, they are typically used after the ureteral stent is placed and the patient has recovered from anesthesia. Other studies have shown no difference in stent symptoms in these two classes of drugs.

The Belladonna and Opium (B&O) suppository is a potent anti-muscarinic medication with narcotic properties. It frequently is used as a second line drug for patients with severe bladder spasms refractory to first line anti-muscarinic and narcotic medications from an indwelling Foley catheter or ureteral stent. It has shown efficacy for Foley catheter discomfort in patients undergoing robotic prostatectomies, but its use in the perioperative period has not been studied for ureteral stent discomfort.

The purpose of this study is to determine if preemptive B&O suppository placement will decrease post-operative pain in patients undergoing ureteral stent placement.

Procedures: The study is a randomized double-blind controlled trial comparing the use of a B&O suppository versus placebo suppository for the preemptive treatment of ureteral stent discomfort. 70 subjects will be recruited from the outpatient urologic clinic under the care of a single surgeon with appropriate informed consent. At the time of recruitment, patients will complete a validated AUA symptom score questionnaire in order to establish baseline symptom scores and urinary bother. Patients will be randomized into a treatment arm or a placebo arm. Those randomized to the treatment arm will receive a single B&O suppository, dose-weight calculated, immediately following patient positioning prior to instrumentation. Those randomized to the other arm will receive a single placebo suppository. The suppository will be administered by the circulating operative nurse and the remainder of the surgical team will be blinded to the study drug. Following treatment and stent placement, all patients will receive standard post-operative pain management (hydrocodone/acetaminophen, docusate, and tamsulosin) with usual discharge instructions.

Subject Population: Primary study population is patients who will receive ureteroscopy with concurrent placement of a ureteral stent. Primary exclusion criteria include age < 18, neurologic deficits of any kind and non-English speaking patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who will receive ureteroscopy with concurrent placement of a ureteral stent.

Exclusion Criteria:

* age < 18,
* neurologic deficits of any kind
* non-English speaking patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Belladonna and Opium (B&O) Suppository: A single belladonna and opium suppository, dose-weight calculated, administered immediately following patient positioning prior to instrumentation. The pharmacologically active ingredients that are present in the belladonna extract consist of atropine and scopolamine. Opium is compound drug that is composed of 20 alkaloids. The principle alkaloid that derives the majority of its effect is its morphine content and acts as a narcotic analgesic by increasing the pain threshold or the magnitude of stimulus required to evoke pain.
  Belladonna and Opium
Period: Overall Study
Arm/Group | Belladonna and Opium (B&O) Suppository | Placebo Suppository
Started | 35 | 36
Completed | 26 | 26
Not Completed | 9 | 10
Not completed — Incomplete questionnaires | 8 | 9
Not completed — Passed stone prior to surgery date | 1 | 0
Not completed — Did not require a ureteral stent | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belladonna and Opium (B&O) Suppository | Placebo Suppository | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13) | 50 (16) | 53 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 18 | 16 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 35 | 36 | 71

OUTCOME MEASURES:

1. Primary Outcome: Global Quality of Life Score on Postoperative Day 1
Description: Global quality of life score as measured by the Ureteral Stent Symptom Questionnaire (USSQ).
  Scale is 1-7 (Lower score indicating better quality of life compared to higher score). 1 = delighted, 2 = pleased, 3 = mostly satisfied, 4 = mixed feelings (about equally satisfied and dissatisfied), 5 = mostly dissatisfied, 6 = unhappy, 7 = terrible
Time Frame: postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belladonna and Opium (B&O) Suppository | Placebo Suppository
Number analyzed (Participants) | 35 | 34
score on a scale | 4.4 (0.6) | 5.4 (1.2)

2. Primary Outcome: Global Quality of Life Score on Postoperative 3
Description: as for outcome 1
Time Frame: postoperative day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Belladonna and Opium (B&O) Suppository | Placebo Suppository
Number analyzed (Participants) | 35 | 34
score on a scale | 4.5 (1.4) | 5.6 (1.3)

3. Secondary Outcome: Number of Participants With Postoperative Complications as a Result of the Use of B&O Suppository
Description: To assess postoperative complications as a result of the use of B&O suppository, including urinary retention.
Time Frame: 14 days post-op
Population: Adverse reactions in the intervention group
Measure: Count of Participants; unit: Participants
Arm/Group | Belladonna and Opium (B&O) Suppository | Placebo Suppository
Number analyzed (Participants) | 35 | 0
Participants | 0 |

4. Secondary Outcome: Number of Participants With Unanticipated Postoperative Visits
Description: Number of postoperative unanticipated visits including nursing visits and ED visits
Time Frame: 14 days post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Belladonna and Opium (B&O) Suppository | Placebo Suppository
Number analyzed (Participants) | 35 | 34
Participants | 3 | 5

5. Secondary Outcome: Measurement of Post-operative Narcotic Use
Description: Measurement of postoperative opiate use using a questionnaire. We will define success as a reduction in postoperative narcotic use by 10% compared to placebo.
Time Frame: 14 days post-op
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Belladonna and Opium (B&O) Suppository | Placebo Suppository
Number analyzed (Participants) | 35 | 34
morphine milligram equivalents | 55 (76) | 65 (79)

ADVERSE EVENTS:
Arm/Group | Belladonna and Opium (B&O) Suppository | Placebo Suppository
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 3/35 | 5/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belladonna and Opium (B&O) Suppository (N=35) | Placebo Suppository (N=34)
Emergency Department visits (General disorders) | 3 (3) | 5 (5) — Postoperative ED visits. Expected is 12-15%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No